CLINICAL TRIAL: NCT00363649
Title: A Randomized Phase II Trial of Interferon + GM-CSF Versus K562/GM-CSF Vaccination in CML Patients Achieving a Complete Cytogenetic Response to Frontline Tyrosine Kinase Inhibitor Therapy
Brief Title: Interferon and GM-CSF Compared With Imatinib Mesylate and Vaccine Therapy in Patients With Chronic Phase CML on a TKI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: J05121; P30CA006973 (NIH)
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-10

CONDITIONS: Leukemia
Keywords: Philadelphia chromosome positive chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — Interferon-alpha; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to Arm A or Arm B and received up to twelve months of protocol therapy. If at any point a participant progressed, relapsed, or had unacceptable toxicity, they could cross over to the other arm. Participants could only cross over once.

ARMS (2):
- Arm A (Experimental): Patients will receive injections of interferon alfa and sargramostim once a day for 6 months. Some patients may receive treatment for up to 1 year. After 1 year, some patients may receive treatment as in arm II.
  Interventions: Biological: Interferon alfa; Biological: Sargramostim
- Arm B (Experimental): Patients will receive an injection of GM-K562 cell vaccine every 3 weeks for at least 6 months. Some patients may receive treatment for up to 1 year. After 1 year, some patients may receive treatment as in arm I. NOTE: Study Arm B is not available to newly accrued and enrolled subjects based on the interim analysis directing all new subjects to the combination of Interferon + sargramostim (Arm A).
  Interventions: Biological: GM-K562 cell vaccine

INTERVENTIONS:
Biological: GM-K562 cell vaccine — Given by injection
  Arms: Arm B
Biological: Interferon alfa — Given by injection
  Arms: Arm A
Biological: Sargramostim — Given by injection
  Other Names: GM-CSF
  Arms: Arm A

SUMMARY:
RATIONALE: Tyrosine kinase inhibitors may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Interferon alfa may interfere with the growth of cancer cells. GM-CSF may help cells that are involved in the body's immune response work better. Vaccines made from a person's cancer cells may help the body build an effective immune response to kill cancer cells.

PURPOSE: This randomized phase II trial is studying tyrosine kinase inhibitors, interferon alfa, and GM-CSF to see how well they work compared to tyrosine kinase inhibitors and vaccine therapy in treating patients with chronic phase chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare clinical response, in terms of 1-year progression-free survival and rate of molecular complete remission, in patients with Philadelphia chromosome-positive chronic myelogenous leukemia (Ph+ CML) in chronic phase who have achieved a complete cytogenetic remission to single-agent tyrosine kinase inhibitor treated with interferon alfa and sargramostim (GM-CSF) vs tyrosine kinase inhibitor and GM-K562 cell vaccine.

Secondary

* Compare time to Ph-negativity by polymerase chain reaction after randomization.
* Compare disease-free survival and percent molecular complete remissions.
* Determine the toxicity of these treatment regimens in these patients.

OUTLINE: This is a multicenter, randomized, crossover, study. Patients are randomized to 1 of 2 treatment arms. The study will be modified based on the results of the planned interim analysis. Individual Study Arms will continue to accrue and treat as indicated by the analysis. The study in its current format will continue should the planned interim analysis indicate both Study Arms remain viable as effective treatments.

All patients continue to receive their standard dose of tyrosine kinase inhibitor in addition to 1 of the following treatment arms:

* Arm I : Patients receive interferon alfa subcutaneously (SC) and GM-CSF SC once daily for 6 months. Patients who achieve a molecular complete remission (CR) (defined as BCR-ABL-negative disease confirmed by 2 PCR assays separated by 1 month) at the end of the 6-month period, discontinue study therapy and are monitored for disease recurrence by blood tests every 4 weeks. Patients who do not achieve a molecular CR (defined as BCR-ABL-positive disease) after completion of the initial 6 months of therapy, receive an additional 6 months of therapy as above. Patients who achieve BCR-ABL-negative disease during the additional 6 months of therapy, discontinue study therapy and are monitored for disease recurrence by blood tests every 4 weeks. Patients who remain BCR-ABL-positive by PCR after an additional 6 months of therapy, are eligible to cross over to arm II.

If at any time after stopping study therapy blood tests show disease recurrence, patients restart tyrosine kinase inhibitor and are eligible to cross over to arm II. Patients are also eligible to cross over to arm II in the presence of unacceptable toxicity.

* Arm II: Patients receive GM-K562 cell vaccine intradermally once every 3 weeks for a minimum of 6 months. Patients with BCR-ABL-negative disease at the end of the 6-month period discontinue study therapy and are monitored for disease recurrence by blood tests every 4 weeks. Patients with BCR-ABL-positive disease after the completion of the initial 6 months of therapy, receive an additional 6 months of therapy as above. Patients who achieve BCR-ABL-negative disease during the additional 6 months of therapy, discontinue study therapy and are monitored every 4 weeks for disease recurrence. Patients who remain BCR-ABL-positive after the additional 6 months of therapy, are eligible to cross over to arm I.

If at any time after stopping study therapy blood tests show disease recurrence, patients restart tyrosine kinase inhibitor and are eligible to cross over to arm I. Patients are also eligible to cross over to arm I in the presence of unacceptable toxicity.

After completion of study therapy, patients are followed periodically for up to 1 year.

As of May 2014, Study Arm B is not available to newly accrued and enrolled subjects based on the interim analysis directing all new subjects to the combination of Interferon + GM-CSF.

PROJECTED ACCRUAL: A total of 56 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic myelogenous leukemia (CML) in chronic phase based on cytogenetic detection of the Philadelphia chromosome and/or detection of the BCR-ABL rearrangement by any of the following molecular methods:

  * Recombinant DNA analysis of the BCR-ABL fusion gene
  * Fluorescence in situ hybridization (FISH)
  * Polymerase chain reaction detection of the BCR-ABL hybrid mRNA
* Documentation of complete cytogenetic response by conventional cytogenetic or FISH analysis while on a stable dose of tyrosine kinase inhibitor
* No other phase of CML

PATIENT CHARACTERISTICS:

* ECG performance status 0-2
* Life expectancy > 24 months
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* Creatinine ≤ 2.0 mg/dL
* Bilirubin ≤ 2.0 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* No other malignancy within the past 5 years except in situ cervical carcinoma or adequately treated nonmelanoma skin cancer
* No other disease requiring long-term corticosteroids or immunosuppressants

PRIOR CONCURRENT THERAPY:

* At least 28 days since prior investigational agents
* No prior bone marrow transplant or other transplant
* No concurrent immunosuppressants (e.g., steroids, cyclosporine, azathioprine, mycophenolate mofetil, sirolimus, or tacrolimus)
* No concurrent hydroxyurea, busulfan, or cytoreductive agents (other than frontline TKI)
* No other concurrent anticancer agents or therapies

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: B. Douglas Smith, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants were screen failures.
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 18 | 16
Crossed Over to Arm B | 9 | 0
Crossed Over to Arm A | 0 | 12
Did Not Cross Over | 2 | 3
Completed | 11 | 15
Not Completed | 7 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 16 | 34
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 43 [23 to 64] | 40 [27 to 64] | 40.5 [23 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 15 | 32
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 15 | 14 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 16 | 34

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Number of patients alive and without disease progression or relapse
Time Frame: 1 year after treatment has been stopped
Population: Crossover participants were not analyzed for this outcome. This is as per the analysis plan written in this protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 18 | 16
Participants | 2 | 0

2. Primary Outcome: Complete Remission Rate
Description: Percentage of patients who achieved molecular remission as defined by polymerase chain reaction negativity.
Time Frame: Up to 18 months
Population: Crossover participants were not analyzed for this outcome. This is as per the analysis plan written in this protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 18 | 16
percentage of participants | 61.1 | 62.5

3. Secondary Outcome: Time to Complete Molecular Remission
Description: Number of months from randomization to molecular remission as defined by polymerase chain reaction negativity.
Time Frame: Up to 27 months
Population: Crossover participants were not analyzed for this outcome. This is as per the analysis plan written in this protocol.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 18 | 16
months | 10 [4.7 to 11.2] | 16.3 [6.9 to 27]

4. Secondary Outcome: Disease-free Survival
Description: Median number of days to progression of disease in participants who stopped all treatment as directed by the protocol.
Time Frame: Up to 8 years
Population: Crossover participants were not analyzed for this outcome. This is as per the analysis plan written in this protocol.
Measure: Median (Full Range); unit: days
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 18 | 16
days | 82 [28 to 2924] | 98 [56 to 116]

5. Secondary Outcome: Early Discontinuation
Description: Number of participants unable to complete protocol-specified treatment due to toxicity.
Time Frame: 1 year
Population: This outcome includes all participants who were either started on an arm or crossed over to an arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 30 | 25
Participants | 10 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Adverse events were collected monthly for up to two years.
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/30 | 0/25
Other Adverse Events (participants affected / at risk) | 30/30 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=30) | Arm B (N=25)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
New malignancy - breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=30) | Arm B (N=25)
Acid reflux (Gastrointestinal disorders) | 1 (1) | 3 (4)
Adenopathy (Immune system disorders) | 5 (5) | 3 (4)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (2)
Alopecia (General disorders) | 4 (4) | 3 (3)
ALT increased (Investigations) | 8 (17) | 3 (5)
Anemia (Investigations) | 6 (12) | 5 (7)
Anorexia (General disorders) | 6 (7) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
AST increased (Investigations) | 7 (10) | 8 (13)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Chills (General disorders) | 2 (2) | 1 (1)
Conjunctivitis (Eye disorders) | 2 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (7)
Dehydration (General disorders) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 2 (2) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 7 (11) | 4 (6)
Dizziness (Nervous system disorders) | 3 (5) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (4)
Edema (Blood and lymphatic system disorders) | 12 (19) | 10 (17)
Fatigue (General disorders) | 19 (32) | 15 (34)
Fever (Infections and infestations) | 5 (9) | 5 (8)
Flu-like symptoms (General disorders) | 18 (28) | 6 (8)
Gastroenteritis (Infections and infestations) | 4 (4) | 5 (5)
Hidradentitis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hyperglycemia (Investigations) | 6 (10) | 5 (6)
Hypertension (Cardiac disorders) | 1 (1) | 3 (3)
Hyperuricemia (Investigations) | 4 (4) | 1 (1)
Hypoalbuminemia (Investigations) | 3 (4) | 0 (0)
Hypocalcemia (Investigations) | 6 (8) | 2 (3)
Hypoglycemia (Investigations) | 1 (1) | 3 (3)
Hypokalemia (Investigations) | 4 (8) | 2 (3)
Indigestion (Gastrointestinal disorders) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 4 (4)
Injection site reaction (Immune system disorders) | 15 (23) | 25 (426)
Infection - sinus (Infections and infestations) | 5 (7) | 9 (12)
Infection - upper respiratory (Infections and infestations) | 3 (3) | 4 (6)
Insomnia (General disorders) | 6 (6) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Leukopenia (Investigations) | 5 (14) | 8 (15)
Lightheadedness (Nervous system disorders) | 0 (0) | 2 (2)
Lymphopenia (Investigations) | 7 (11) | 3 (4)
Malaise (General disorders) | 1 (1) | 1 (1)
Menstrual cycle changes (Reproductive system and breast disorders) | 4 (4) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (9) | 3 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 7 (9)
Nasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4)
Nausea (Gastrointestinal disorders) | 11 (11) | 5 (5)
Night sweats (General disorders) | 3 (3) | 1 (1)
Pain - abdomen (Gastrointestinal disorders) | 3 (4) | 1 (2)
Pain - back (Musculoskeletal and connective tissue disorders) | 5 (7) | 0 (0)
Pain - bone (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (8)
Pain - ear (General disorders) | 2 (2) | 0 (0)
Pain - generalized (General disorders) | 4 (4) | 3 (3)
Pain - head (General disorders) | 8 (12) | 8 (19)
Pain - leg (Musculoskeletal and connective tissue disorders) | 6 (8) | 0 (0)
Pain - throat (Gastrointestinal disorders) | 4 (4) | 7 (9)
Pigmentation changes (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Post-nasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Eye swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 10 (12) | 6 (6)
Rigors (General disorders) | 2 (5) | 0 (0)
Seasonal allergies (Immune system disorders) | 1 (1) | 1 (1)
Ankle sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Investigations) | 4 (9) | 2 (4)
Viral infection (Infections and infestations) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (4)
Watery eyes (Eye disorders) | 2 (2) | 2 (3)
Weakness (Nervous system disorders) | 1 (1) | 1 (1)
Weight gain (General disorders) | 1 (1) | 2 (2)
Xerosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Xerostomia (Gastrointestinal disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT00363649/Prot_SAP_000.pdf